CLINICAL TRIAL: NCT05697744
Title: Evaluation of Vidiac Scores of Obese and Morbid Obese Patients Intubated by Videolaryngoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, aysun postaci, Ankara City Hospital Bilkent, Ankara City Hospital Bilkent
Other Study IDs: E2-23-3157
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Vidiac Score; Videolaryngoscopy; Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese: Vidiac score Mallampati score upper lip bite test Thyromental distance Mandible ramus length Mouth opening distance
  Interventions: Diagnostic Test: Vidiac Score
- Morbid obese: Vidiac score Mallampati score upper lip bite test Thyromental distance Mandible ramus length Mouth opening distance
  Interventions: Diagnostic Test: Vidiac Score

INTERVENTIONS:
Diagnostic Test: Vidiac Score — Vidiac score is a scoring system created according to the visibility of laryngeal structures under videolarnyngoscopy in patients with expected difficult intubation.

SUMMARY:
The aim of the study was to observe the vidiac score values of only patients with obesity as a risk factor for difficult intubation. Secondly, it was aimed to evaluate the number of intubation attempts and intubation time, vidiac scores between obese and morbid obese patients and to reveal the differences, if any.

ELIGIBILITY:
Inclusion Criteria:

* All obese and morbidly obese patients to be operated under general anesthesia and endotracheal intubation

Exclusion Criteria:

1. under 18 years old
2. The patient's refusal
3. Difficult airway story before
4. Congenital or previous airway anatomical disorder
5. Patients who have undergone airway surgery
6. Patients with a mass in the head and neck region
7. Body mass ındex < 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients to be operated under general anesthesia and endotracheal intubation
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
vidiac score | during entubation
  Vidiac score is a scoring system created according to the visibility of laryngeal structures under videoingoscopy in patients with expected difficult intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Postacı, Assoc. Prof, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided